CLINICAL TRIAL: NCT03571204
Title: An Exploratory Study of Combination Therapy With 3BNC117 and 10-1074 in HIV-Infected Individuals
Brief Title: Combination Therapy With 3BNC117 and 10-1074 in HIV-Infected Individuals
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Coronavirus 2019 (COVID-19) pandemic
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 180115; 18-I-0115 (Other: NIHCC)
Record Dates: First submitted 2018-06-22; First posted 2018-06-27 (Actual); Results first posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2021-03

CONDITIONS: HIV
Keywords: Treatment Interruption; Neutralizing Monoclonal Antibody

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: ART prior to 3BNC117 + 10-1074 in HIV-1 subject (Active Comparator): Subjects who began anti-retroviral therapy (ART) during primary HIV-1 infection within 12 weeks of diagnosis. ART was stopped after study day 3 and were given 3BNC117 and 10-1074 intravenously. Both 3BNC117 and 10-1074 were administered at 30 mg/kg dose level in separate bags of 250 mL normal saline in sequential administration. Subjects received 8 infusions of 3BNC117 and 10-1074 at weeks 0, 2, 4, 8, 12, 16, 20, and 24. The total duration of therapy was 24 weeks.
  Interventions: Biological: 3BNC117 and 10-1074
- Group 1: ART prior to placebo treatment in HIV-1 subject (Placebo Comparator): Subjects who began anti-retroviral therapy (ART) during primary HIV-1 infection within 12 weeks of diagnosis. ART was stopped after study day 3 and were given normal saline intravenously. Subjects received two separate bags of 250 mL normal saline in sequential administration. Subjects received 8 infusions at weeks 0, 2, 4, 8, 12, 16, 20, and 24. The total duration of therapy was 24 weeks.
  Interventions: Biological: Placebo
- Group 2: 3BNC117 + 10-1074 in HIV-1 subject (Experimental): Subjects who were not on anti-retroviral therapy (ART) during primary HIV-1 infection within the past 2 years. Subjects were given 3BNC117 and 10-1074 intravenously. Both 3BNC117 and 10-1074 were administered at 30 mg/kg dose level in separate bags of 250 mL normal saline in sequential administration. Subjects received 8 infusions of 3BNC117 and 10-1074 at weeks 0, 2, 4, 8, 12, 16, 20, and 24. The total duration of therapy was 24 weeks.
  Interventions: Biological: 3BNC117 and 10-1074

INTERVENTIONS:
Biological: 3BNC117 and 10-1074 — Both 3BNC117 and 10-1074 administered intravenously at 30 mg/kg dose level in 250 ml normal saline for 8 infusions at weeks 0, 2, 4, 8, 12, 16, 20, and 24. The two antibodies will be mixed in separate bags of saline for sequential administration.
  Arms: Group 1: ART prior to 3BNC117 + 10-1074 in HIV-1 subject; Group 2: 3BNC117 + 10-1074 in HIV-1 subject
Biological: Placebo — Placebo is two separate bags of 250 ml normal saline administered intravenously for 8 infusions at weeks 0, 2, 4, 8, 12, 16, 20, and 24. The two separate bags of placebo are administered sequentially.
  Arms: Group 1: ART prior to placebo treatment in HIV-1 subject

SUMMARY:
Background:

Human immunodeficiency virus (HIV) affects the immune system. The main function of the immune system is protect you from infections and other diseases such as cancer. HIV attacks and cripples the immune system making people more susceptible to a variety of infections and cancers. Currently, the standard treatment for HIV infection is a daily administration of anti-HIV drugs. These drugs are called combination antiretroviral therapy (ART). ART is very effective at suppressing HIV, but does not cure HIV infection. ART must be taken continuously for life to be effective. ART can stop being effective if not taken correctly and can cause permanent side effects. Researchers want to see if two new products can control HIV infection without the use of ART. The products are the antibodies 3BNC117 and 10-1074.

Objective:

To see if 3BNC117 and 10-1074 are safe and can control HIV levels in the blood of people who are not taking ART or people who stop taking their ART during the study. .

Eligibility:

Adults ages 18-65 with HIV who are:

* on ART and willing to stop treatment for at least 28 weeks
* OR not taking ART with low levels of HIV in the blood

Design:

Participants will be screened with a physical exam, medical history, and blood, heart, and urine tests.

Participants will get the 2 study products or salt water (placebo). A thin tube will be placed in an arm vein. Each product will be given directly into the vein for about 1 hour.

To help collect blood cells to study in the laboratory, participants may have a procedure known as leukapheresis in which blood will be removed through a needle in the arm. Some of the white blood cells will be separated from the blood and used for research studies to see how 3BNC117 and 10-1074 effects HIV and the immune system. The rest of the blood will be returned to the person through another needle in the arm.

Participants will have 18 study visits over 28 weeks. They will repeat some screening tests. They may have leukapheresis again.

At 8 study visits, participants will get the study products or placebo.

All participants will be followed for at least 24 weeks after their last dose of the study infusions. Participants who are in the Group that stops ART will be monitored closely to make sure the levels of virus in their blood do not go to high. If at any time during this the study a person develops HIV-related symptoms, or if the viral levels go up to high levels for more than 4 weeks, ART will be restarted and no further infusions of 3BNC117 and 10-1074 will be given.

...

DETAILED DESCRIPTION:
Recent advances in antibody cloning technologies have led to the discovery of a number of highly potent and HIV-specific broadly neutralizing monoclonal antibodies (bNAbs) from B cells of HIV-infected individuals. It has been shown that certain bNAbs can prevent acquisition of the virus, suppress viral replication, delay and/or prevent plasma viral rebound following treatment interruption in Simian Immunodeficiency virus (SIV)-infected animals and block cell-to-cell transmission of laboratory-adapted HIV in vitro. In light of these encouraging outcomes, a number of clinical trials have been conducted in recent years in order to explore the feasibility of achieving sustained virologic suppression using a single bNAb in HIV-infected individuals following analytical treatment interruption (ATI). Despite the fact that repeated administration of a single bNAb was safe and well-tolerated, the vast majority of study subjects experienced plasma viral rebound following ATI, clearly demonstrating that successful passive immunotherapy will require different approach, including the use of a combination of 2 or more bNAbs to achieve extended periods of virologic suppression.

Given a major emphasis on current HIV research lies in the possibility of achieving ART-free virologic remission, it is of great interest to investigate whether a combination of potent HIV- specific bNAbs, such as 3BNC117 and 10-1074, can prevent plasma viral rebound in infected individuals upon discontinuation of ART or suppress viral replication in subjects who are not taking ART.

ELIGIBILITY:
* INCLUSION CRITERIA:

General Inclusion Criteria for both Groups:

1. Age 18-65 years old.
2. HIV-1 infection and clinically stable.
3. General good health and has an identified primary health care provider for medical management of HIV infection and is willing to maintain a relationship with a primary health care provider for medical management of HIV infection while participating in the study.
4. Cluster of differentiation 4 (CD4)+ T cell count >450 cells/mm(3) at screening.
5. Laboratory values within pre-defined limits at screening:

   1. Absolute neutrophil count >1,000/mm(3).
   2. Hemoglobin levels >10.0 g/dL for men and >9.0 g/dL for women.
   3. Platelet count >100,000/mm(3).
   4. Estimated or a measured glomerular filtration rate >60 mL/min/1.73m(2) as determined by the National Institutes of Health (NIH) Clinical Center laboratory.
   5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels of <2.5 times upper limit of normal (ULN), direct bilirubin within the normal range for the NIH Clinical Center laboratory.
6. Willingness to have samples stored for future research.

   Inclusion criteria specific for Group 1:
7. Institution of ART within 12 weeks of being diagnosed with primary HIV-1 infection
8. Primary HIV-1 infection is defined as meeting at least one of the following criteria:

   1. Detectable plasma HIV-1 RNA levels of >2000 copies/mL with a negative result from an HIV-1 enzyme immunoassays (EIA), or
   2. Positive result from an HIV-1 EIA with a negative or indeterminate result from an HIV-1 western blot or another confirmatory antibody test that subsequently evolves to a confirmed positive result, or
   3. Negative result from an HIV-1 EIA within the past 4 months and HIV-1 RNA levels of >400,000 copies/mL, in the setting of a potential exposure to HIV-1.
   4. Negative result from an HIV-1 EIA within 6 months prior to a positive result from an HIV-1 EIA and an HIV-1 western blot or another confirmatory antibody test.
   5. Presence of low level of HIV antibodies as determined by having a positive EIA or a positive Western blot with a non-reactive detuned EIA according to a serologic testing algorithm for recent infection.
9. Documentation of continuous ART treatment with suppression of plasma viral level below the limit of detection for greater than or equal to 1 years. Individuals with blips (i.e., detectable viral levels on ART) prior to screening may be included provided they satisfy the following criteria:

   1. The blips are <400 copies/mL, and
   2. Succeeding viral levels return to levels below the limit of detection on subsequent testing.
10. Willingness to undergo ATI
11. Willingness for both male and female subjects to agree to use barrier protection methods or abstinence during the ATI phase of the study to decrease the risk of HIV transmission.

    Inclusion criteria specific for Group 2:
12. No ART within 24 months of screening.
13. HIV plasma viremia between 200 and 5,000 copies/mL at screening AND at least two documented viral level greater than or equal to 200 copies/mL in the 12 months prior to screening.

At the screening visit, subjects considering enrollment in Group 2 will be advised that current guidelines recommend treatment of all individuals with HIV infection regardless of viral levels and CD4 counts.

Reproductive Risks

Contraception: The effects of 3BNC117 and 10-1074 on the developing human fetus are unknown. For this reason, men and women of childbearing potential must agree to use adequate pregnancy prevention. This includes the use an effective method of contraception (i.e. condom with spermicide, diaphragm with spermicide, hormone-eluting intrauterine device (IUD), hormone-based contraceptive with condom) for the study duration. Subjects should also agree to use a male or female condom while off ART. Pregnancy prevention must be practiced continuously for the duration of study participation. Females of childbearing-age must have a negative pregnancy test result prior to receiving each infusion of 3BNC117/10-1074. During the course of the study, if a female subject, or the partner of a male subject suspects or in fact becomes pregnant, the effected subject should inform the study staff immediately, as well as the woman s primary care physician.

EXCLUSION CRITERIA:

1. Chronic hepatitis B, as evidenced by a positive test for hepatitis B surface antigen

   (HBsAg), or chronic hepatitis C virus (HCV) infection, as evidenced by a positive test for HCV RNA. Subjects with a positive test for HCV antibody and a negative test for HCV RNA are eligible.
2. HIV immunotherapy or vaccine(s) received within 1 year prior to screening.
3. Any licensed or experimental non-HIV vaccination (e.g., hepatitis B, influenza, pneumococcal polysaccharide) received within 2 weeks prior to study enrollment.
4. Receipt of other investigational study agent within 28 days of enrollment.
5. Any active malignancy that may require systemic chemotherapy or radiation therapy.
6. Systemic immunosuppressive medications received within 3 months prior to enrollment (Not excluded: [1] corticosteroid nasal spray or inhaler; [2] topical corticosteroids for mild, uncomplicated dermatitis; or [3] oral/parenteral corticosteroids administered for non-chronic conditions not expected to recur [length of therapy less than or equal to10 days, with completion in greater than or equal to 30 days prior to enrollment]).
7. History or other clinical evidence of:

   1. Significant or unstable cardiac or cerebrovascular disease (e.g., angina, congestive heart failure, recent stroke or myocardial infarction).
   2. Severe illness, malignancy, immunodeficiency other than HIV, or any other condition that, in the opinion of the investigator, would make the subject unsuitable for the study.
8. Active drug or alcohol use or any other pattern of behavior that, in the opinion of the investigator, would interfere with adherence to study requirements.
9. Pregnancy or breast-feeding at time of screening.
10. Documented multiclass antiretroviral drug resistance that, in the judgment of the investigator, would pose a risk of virologic failure should additional mutations develop during the study (Group 1 only).

Co-enrollment Guidelines: Co-enrollment in other trials is restricted to observational studies or those evaluating the use of a licensed medication and is subject to approval of the principal investigator (PI).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Sneller, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Caskey M, Klein F, Lorenzi JC, Seaman MS, West AP Jr, Buckley N, Kremer G, Nogueira L, Braunschweig M, Scheid JF, Horwitz JA, Shimeliovich I, Ben-Avraham S, Witmer-Pack M, Platten M, Lehmann C, Burke LA, Hawthorne T, Gorelick RJ, Walker BD, Keler T, Gulick RM, Fatkenheuer G, Schlesinger SJ, Nussenzweig MC. Viraemia suppressed in HIV-1-infected humans by broadly neutralizing antibody 3BNC117. Nature. 2015 Jun 25;522(7557):487-91. doi: 10.1038/nature14411. Epub 2015 Apr 8. PMID 25855300
- [Background] Caskey M, Schoofs T, Gruell H, Settler A, Karagounis T, Kreider EF, Murrell B, Pfeifer N, Nogueira L, Oliveira TY, Learn GH, Cohen YZ, Lehmann C, Gillor D, Shimeliovich I, Unson-O'Brien C, Weiland D, Robles A, Kummerle T, Wyen C, Levin R, Witmer-Pack M, Eren K, Ignacio C, Kiss S, West AP Jr, Mouquet H, Zingman BS, Gulick RM, Keler T, Bjorkman PJ, Seaman MS, Hahn BH, Fatkenheuer G, Schlesinger SJ, Nussenzweig MC, Klein F. Antibody 10-1074 suppresses viremia in HIV-1-infected individuals. Nat Med. 2017 Feb;23(2):185-191. doi: 10.1038/nm.4268. Epub 2017 Jan 16. PMID 28092665
- [Background] Bar KJ, Sneller MC, Harrison LJ, Justement JS, Overton ET, Petrone ME, Salantes DB, Seamon CA, Scheinfeld B, Kwan RW, Learn GH, Proschan MA, Kreider EF, Blazkova J, Bardsley M, Refsland EW, Messer M, Clarridge KE, Tustin NB, Madden PJ, Oden K, O'Dell SJ, Jarocki B, Shiakolas AR, Tressler RL, Doria-Rose NA, Bailer RT, Ledgerwood JE, Capparelli EV, Lynch RM, Graham BS, Moir S, Koup RA, Mascola JR, Hoxie JA, Fauci AS, Tebas P, Chun TW. Effect of HIV Antibody VRC01 on Viral Rebound after Treatment Interruption. N Engl J Med. 2016 Nov 24;375(21):2037-2050. doi: 10.1056/NEJMoa1608243. Epub 2016 Nov 9. PMID 27959728
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-I-0115.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: of 27 participants consented, 6 participants were screen failure so did not start the actual study.
Period: Overall Study
Arm/Group | Group 1: ART Prior to 3BNC117 + 10-1074 in HIV-1 Subject | Group 1: ART Prior to Placebo Treatment in HIV-1 Subject | Group 2: 3BNC117 + 10-1074 in HIV-1 Subject
Started | 8 | 8 | 5
Completed | 7 | 6 | 5
Not Completed | 1 | 2 | 0
Not completed — Stopped due to COVID-19 pandemic | 1 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Group 2 ART naiive
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: ART Prior to 3BNC117 + 10-1074 in HIV-1 Subject | Group 1: ART Prior to Placebo Treatment in HIV-1 Subject | Group 2: 3BNC117 + 10-1074 in HIV-1 Subject | Total
Number analyzed (Participants) | 8 | 8 | 5 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 5 | 21
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 8 | 8 | 5 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 7 | 6 | 5 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 4 | 7 | 3 | 14
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Participants With Grade 3 or Higher Adverse Events
Description: Participants with grade 3 or higher adverse events (AE), including serious adverse advents. AE severity was graded according to the Division of Aids Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.1, July, 2017
Time Frame: 29 months
Population: Participants who started the study
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ART Prior to 3BNC117 + 10-1074 in HIV-1 Subject | Group 1: ART Prior to Placebo Treatment in HIV-1 Subject | Group 2: 3BNC117 + 10-1074 in HIV-1 Subject
Number analyzed (Participants) | 8 | 8 | 5
Participants | 0 | 0 | 0

2. Secondary Outcome: Participants Who Experienced Rebound of Plasma Viremia
Description: Difference between the treatment and placebo arms in the number of participants who experienced rebound of plasma viremia and met criteria to restart ART prior to study week 28.
Time Frame: 28 weeks
Population: Participants who initiated anti-retroviral treatment interruption (ATI). Two participants did not participate in ATI. One participant deviated from the protocol and was lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ART Prior to 3BNC117 + 10-1074 in HIV-1 Subject | Group 1: ART Prior to Placebo Treatment in HIV-1 Subject
Number analyzed (Participants) | 7 | 7
Participants | 0 | 6

3. Secondary Outcome: Participants Who Achieved Suppression of Viremia
Description: Participants who achieved suppression of viremia to <40 copies/ml by study week 28
Time Frame: 28 weeks
Population: Participants who started intravenous infusion therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: 3BNC117 + 10-1074 in HIV-1 Subject
Number analyzed (Participants) | 5
Participants | 2

ADVERSE EVENTS:
Time Frame: 29 months
Arm/Group | Group 1: ART Prior to 3BNC117 + 10-1074 in HIV-1 Subject | Group 1: ART Prior to Placebo Treatment in HIV-1 Subject | Group 2: 3BNC117 + 10-1074 in HIV-1 Subject
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 1/5
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: ART Prior to 3BNC117 + 10-1074 in HIV-1 Subject (N=8) | Group 1: ART Prior to Placebo Treatment in HIV-1 Subject (N=8) | Group 2: 3BNC117 + 10-1074 in HIV-1 Subject (N=5)
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: ART Prior to 3BNC117 + 10-1074 in HIV-1 Subject (N=8) | Group 1: ART Prior to Placebo Treatment in HIV-1 Subject (N=8) | Group 2: 3BNC117 + 10-1074 in HIV-1 Subject (N=5)
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 1
Chalazion (Eye disorders) | 0 | 1 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Tooth disorder (Gastrointestinal disorders) | 0 | 0 | 1
Chills (General disorders) | 2 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Infusion site extravasation (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Abscess oral (Infections and infestations) | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Chlamydial infection (Infections and infestations) | 1 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 3 | 2 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 0
Amylase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 0
Blood bicarbonate decreased (Investigations) | 0 | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Blood calcium decreased (Investigations) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 0
Blood glucose increased (Investigations) | 6 | 1 | 3
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0
Blood phosphorus decreased (Investigations) | 4 | 2 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 2
Haemoglobin decreased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due the the COVID-19 pandemic. The pre-defined samples size of 30 participants (15 per arm) for Group 1 was not not reached prior to closing the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/04/NCT03571204/Prot_SAP_000.pdf